CLINICAL TRIAL: NCT00951990
Title: A Multicenter Randomized Controlled Trail of Ergometer Cycling After Hip and Knee Replacement Surgery
Brief Title: Ergometer Cycling After Replacement of the Hip or Knee Joint
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Verein zur Förderung der Rehabilitationsforschung in Schleswig-Holstein (Other)
Collaborators: Verein zur Förderung der Erforschung und Bekämpfung rheumatischer Erkrankungen Bad Bramstedt e.V (Other); Landesversicherungsanstalt Schleswig-Holstein (Unknown); Landesversicherungsanstalt Freie und Hansestadt Hamburg (Unknown); Deutsche Arthrose-Hilfe (Other)
Responsible Party: Thoralf R Liebs, University of Schleswig-Holstein Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: vffr-37
Record Dates: First submitted 2009-08-02; First posted 2009-08-04 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Ergometer Cycling — Ergometer Cycling under the guidance of a physical therapist after the second postoperative week. These training sessions were scheduled to be performed three times a week for a time period of at least three weeks. The resistance of the ergometer was set to a minimum (for example 30 Watts). Physical therapists were informed to pay special attention, that the height of the saddle is set so that the forefoot reaches the pedal with the knee in extension.
Behavioral: No ergometer cycling — Patients of the no ergometer cycling group did not receive any ergometer cycling after surgery

SUMMARY:
Despite the widespread use of hip and knee replacement surgery, there is a considerable lack of consensus regarding postoperative treatment and rehabilitation, mostly because of the lack of well-designed studies testing the efficacy and effectiveness of such practices.

In particular there are no recommendations regarding the use of ergometer cycling after hip or knee replacement surgery.

Therefore the investigators initiated a multicenter controlled clinical trial evaluating the effect of ergometer cycling versus no ergometer cycling after hip or knee replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is about to receive unilateral hip or knee replacement surgery on an elective basis of diagnosis of osteoarthritis or femoral head necrosis

Exclusion Criteria:

* A history of septic arthritis
* Hip fracture
* Intraoperative complications
* History of implant surgery on the joint to be operated on
* Rheumatoid arthritis
* Amputations
* Inability of complete the questionnaires because of cognitive or language difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 457 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
WOMAC Physical Function | 3 months to 24 months

SECONDARY OUTCOMES:
WOMAC Pain and Stiffness | 3 months to 24 months
SF-36 | 3 months to 24 months
Patient satisfaction | 3 months to 24 months
Lequesne Hip or Knee Score | 3 months to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Hassenpflug, PhD, Study Chair — University of Schleswig-Holstein Medical Center, Department of Orthopedic Surgery, Kiel Campus, 24105 Kiel, Germany
Locations (5):
- Germany (5):
  - Rheumaklinik Bad Bramstedt, Department of Orthopedic Surgery, Bad Bramstedt
  - Ostseeklinik Damp, Department I of Orthopedic Surgery, Damp
  - University of Schleswig-Holstein Medical Center, Department of Orthopedic Surgery, Kiel
  - University of Schleswig-Holstein Medical Center, Lübeck Campus, Lübeck
  - Wedel Hospital, Department of Surgery, Wedel

REFERENCES:
- [Background] Liebs TR, Nasser L, Herzberg W, Ruther W, Hassenpflug J. The influence of femoral offset on health-related quality of life after total hip replacement. Bone Joint J. 2014 Jan;96-B(1):36-42. doi: 10.1302/0301-620X.96B1.31530. PMID 24395308
- [Background] Liebs TR, Herzberg W, Gluth J, Ruther W, Haasters J, Russlies M, Hassenpflug J. Using the patient's perspective to develop function short forms specific to total hip and knee replacement based on WOMAC function items. Bone Joint J. 2013 Feb;95-B(2):239-43. doi: 10.1302/0301-620X.95B2.28383. PMID 23365035
- [Background] Liebs TR, Herzberg W, Roth-Kroeger AM, Ruther W, Hassenpflug J. Women recover faster than men after standard knee arthroplasty. Clin Orthop Relat Res. 2011 Oct;469(10):2855-65. doi: 10.1007/s11999-011-1921-z. Epub 2011 Jun 23. PMID 21698485
- [Background] Liebs TR, Kloos SA, Herzberg W, Ruther W, Hassenpflug J. The significance of an asymmetric extension gap on routine radiographs after total knee replacement: A new sign and its clinical significance. Bone Joint J. 2013 Apr;95-B(4):472-7. doi: 10.1302/0301-620X.95B4.31080. PMID 23539698
- [Result] Liebs TR, Herzberg W, Ruther W, Haasters J, Russlies M, Hassenpflug J. Ergometer cycling after hip or knee replacement surgery: a randomized controlled trial. J Bone Joint Surg Am. 2010 Apr;92(4):814-22. doi: 10.2106/JBJS.H.01359. PMID 20360503
- [Result] Liebs TR, Herzberg W, Ruther W, Russlies M, Hassenpflug J; Multicenter Arthroplasty Aftercare Project, MAAP. Quality-Adjusted Life Years Gained by Hip and Knee Replacement Surgery and Its Aftercare. Arch Phys Med Rehabil. 2016 May;97(5):691-700. doi: 10.1016/j.apmr.2015.12.021. Epub 2016 Jan 11. PMID 26792619